CLINICAL TRIAL: NCT03953664
Title: The Effects of Three Different Modalities of Exercise Training (Aerobic, Strength, Aerobic-strength) on Psychological and Physiological Correlates in Schizophrenia: a Randomized Clinical Trial
Brief Title: The Effects of Three Different Modalities of Exercise in Patients With Schizophrenia
Acronym: E-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-22
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental-Strength training (Experimental): Each session lass 60 minutes, during which time 20 minutes are allocated for warming up and cooling down (stretching) and 40 minutes are allocated to strength training exercise involving the major muscle groups.
  Interventions: Other: Experimental-Exercise training
- Experimental-Aerobic training (Experimental): Each session lass 60 minutes, during which time 20 minutes are allocated for warming up and cooling down (stretching) and 40 minutes are allocated to brisk walking.
  Interventions: Other: Experimental-Exercise training
- Experimental-Strength/Aerobic training (Experimental): Each session lass 60 minutes, during which time 20 minutes are allocated for warming up and cooling down (stretching), 15 minutes are allocated to brisk walking and 25 minutes are allocated to strength training involving the major muscle groups.
  Interventions: Other: Experimental-Exercise training

INTERVENTIONS:
Other: Experimental-Exercise training — Each session lass 60 minutes, during which time 20 minutes are allocated for warming up and cooling down (stretching) and 40 minutes are allocated to strength or/and aerobic training exercises.

SUMMARY:
Exercise has been shown to improve health in patients with schizophrenia. However, it remains unclear which modality of exercise reports better benefits.

Aim: To compare the effects of different modalities of exercise training on psychological and physiological variables in schizophrenia.

DETAILED DESCRIPTION:
Exercise has been shown to improve psychological, physiological, and biological correlates in patients with schizophrenia. However, it remains unclear which modality of exercise reports better health benefits.

Aim: To compare the effects of three different modalities of exercise (aerobic, strength, aerobic-strength) on psychological and physiological variables in patients with schizophrenia.

Design: Randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia
* Age between 18-65 years

Exclusion Criteria:

* Patients with other mental diseases
* Patients with mental disabilities
* Patients who present motor or behavioral pathologies that prevent the realization of the exercise training.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 16 weeks
  Symptoms of schizophrenia are measured according to the subscale scores and total score on the PANSS which consists of 30 items scored from 1 (Absent) to 7 (Extreme). Scores range from 30 to 210, with higher scores indicating more symptoms.

SECONDARY OUTCOMES:
World Health Organization Quality of Life-Short version (WHOQOL-BREF) | 16 weeks
  The WHOQOL-BREF contains 24 questions covering 4 domains plus two questions related to overall quality of life and satisfaction with health. Highes scores represent higher quality of life.
Body Mass Index (BMI) | 16 weeks
  The BMI is defined as the body mass divided by the square of the body height.

CONTACTS AND LOCATIONS:
Overall Officials: JF Lisón, PhD, Study Director — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Moncada, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data will be available to other researchers.
Supporting Information: Study Protocol
Time Frame: Inmediately following publication.